CLINICAL TRIAL: NCT01559584
Title: A Clinical and Immunological Study of Phototoxic Doses of Ultraviolet A for Treatment of Alopecia Areata: A Randomized Controlled Clinical Trial
Brief Title: Phototoxic Doses of Ultraviolet A for Treatment of Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda Mohamed Rasheed, Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Phototoxic UVA in alopecia
Record Dates: First submitted 2012-03-12; First posted 2012-03-21 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Alopecia Areata
Keywords: Alopecia; Areata; Phototherapy; Phototoxic; Ultraviolet A; Randomized controlled trial; Interferon gamma; Transforming growth factor beta-1; Insulin like growth factor-1
MeSH Terms: conditions — Alopecia Areata; Alopecia; Camurati-Engelmann Syndrome | interventions — PUVA Therapy; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phototherapeutic (Experimental): 0.5% solution of 8-methoxypsoralen (MOP) will be applied 20 minutes before UVA exposure (315-400nm).
  UVA sessions will be carried out twice weekly aiming to achieve a phototoxic reaction, in the form of erythema and vesiculation. Once a phototoxic reaction will be achieved, the patient will be asked to rest until the reaction subsides and then resume the phototherapy sessions.
  Interventions: Radiation: ultraviolet A (UVA)
- Conventional therapy (Active Comparator): One monthly injections of intralesional potent corticosteroids
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Radiation: ultraviolet A (UVA) — 0.5% solution of 8-methoxypsoralen (MOP) will be applied 20 minutes before UVA exposure (315-400nm).
  UVA sessions will be carried out twice weekly aiming to achieve a phototoxic reaction, in the form of erythema and vesiculation. Once a phototoxic reaction will be achieved, the patient will be asked to rest until the reaction subsides and then resume the phototherapy sessions.
  Arms: Phototherapeutic
Drug: Triamcinolone Acetonide — One monthly injections of intralesional triamcinolone acetonide
  Arms: Conventional therapy

SUMMARY:
Alopecia areata (AA) is a disease of the hair follicles with multifactorial etiology and a strong component of autoimmune origin. It is characterized by non-scarring hair loss on the scalp or any hair-bearing surface.

Various therapeutic agents have been described for the treatment of AA, but none are curative or preventive. The aim of AA treatment is to suppress the activity of the disease. Phototherapy in the form of topical psoralen and ultraviolet A (PUVA) has been a well documented therapy for AA since 1978.

A more recent technique of topical PUVA, namely phototoxic PUVA, has been adopted in two previous studies. Sessions were carried out once every 3 months, and a higher efficacy with more encouraging response rates in comparison to the conventional PUVA therapy has been documented. This assumed upper hand over the conventional PUVA might be due to increasing the amount of UV reaching the hair follicle cells and the surrounding inflammatory cells. Also it has been suggested that it might play a role as a powerful initiating agent of suppression through direct action at the DNA level. However, still the exact effect of this treatment has not been fully clarified.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with alopecia areata, patchy type (max 3 patches not exceeding 50% of the scalp surface area) of more than 2 months duration.
* Age: 12 years and above

Exclusion Criteria:

* Age: Less than 12 years old.
* Affection of more than 50% of the scalp area
* Diagnosis or history of local dermatological disease in the scalp apart from AA such as eczema, seborrheic dermatitis, psoriasis,..
* Any present / past history of dermatological disease with a potential for koebnerization such as psoriasis, vitiligo.
* Diagnosis or history of any contraindication to receiving phototherapy such as malignancy, systemic lupus
* Dermoscopic evaluation revealing absence of any signs of presence of hair follicles.
* Any psychiatric illness or psychological state impairing future compliance or influencing expectations of the patient.
* Patients with AA totalis or Ophiasis

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Treatment success | After six months from onset of treatment
  Treatment success defined as effective sustained growth of hair in more than 80% of the affected area at the EOS. Clinical assessment will be performed by one non-blinded, and two blinded investigators.

SECONDARY OUTCOMES:
Tissue cytokines response to therapy | At early hair regrowth, but no later than three months of treatment onset, in case of failed hair regrowth
  Explanation at the molecular level of possible mechanisms underlying hair regrowth in responsive patients by assessing tissue levels of IFN-γ, IGF-1 and TGF-Beta1
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | After six months from onset of treatment
  Adverse events will be meticulously monitored all through the study, including hypo/hyper pigmentation, severe erythema, itching or burning sensation.

CONTACTS AND LOCATIONS:
Overall Officials: Hoda M Rasheed, MD, Study Chair — Cairo University; Nermin El-Eishi, MD, Principal Investigator — Cairo University; Vanessa G Hafez, MD, Principal Investigator — Cairo University; Solwan I Elsamanoudy, MBBCh, Principal Investigator — Cairo University; Rehab A Hegazy, MD, Principal Investigator — Cairo University; Olfat G Shaker, MD, Principal Investigator — Cairo University
Locations (1):
- Dermatology department - faculty of medicine- Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] El-Mofty M, Rasheed H, El-Eishy N, Hegazy RA, Hafez V, Shaker O, El-Samanoudy SI. A clinical and immunological study of phototoxic regimen of ultraviolet A for treatment of alopecia areata: a randomized controlled clinical trial. J Dermatolog Treat. 2019 Sep;30(6):582-587. doi: 10.1080/09546634.2018.1543847. Epub 2019 Jan 8. PMID 30411986